CLINICAL TRIAL: NCT03007849
Title: A Pilot Study of Fecal Microbiome and Neutrophil Cellular Adhesion Molecules in Patients With Sickle Cell Disease (SCD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Seah Lim, DIRECTOR OF HEMATOLOGY, Rhode Island Hospital
Other Study IDs: 021316
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with sickle cell disease often develop painful crisis without any obvious reasons. Some patients are more likely to develop this complication than others. It is now clear that painful crisis only occurs when sickled red blood cells stick to white blood cells that have been activated, usually by inflammation or infections. A recent study in mice with sickle cell disease showed that the use of long term antibiotics could reduce the number of activated white blood cells and reduce death of the mice during sickle cell crisis.

The investigators believe that sickle cell patients who develop frequent painful crisis may have a different pattern of bacteria in their intestine when compared to those whose painful crisis occurs infrequently. In this study, the investigators propose to study sickle cell subject's blood to determine how many activated white blood cells he/she have. The investigators will also examine his/her stool to compare the bacteria in his/her stool to those other sickle cell patients. The investigators will then investigate whether or not the results from the blood and stool tests correlate with how frequently the patient develops painful crisis.

The investigators will examine the patients' medical records to find out how many times they have been admitted to the hospital for sickle cell crisis in the last 12 months. The investigators will also obtain information on the following: their age, their sex, whether they are taking hydroxyurea or Penicillin, when they last had a transfusion or exchange transfusion therapy and painful crisis needing hospital admission, whether they have received any antibiotics (other than Penicillin) in the last 4 weeks, and whether they are experiencing a painful crisis at the time that they enter the study. The investigators will obtain, from their previous laboratory results, their levels of hemoglobin F and markers of inflammation. The investigators will check their hemoglobin F level if they have not already had this tested.

The investigators expect to enroll 50 subjects into this study at Rhode Island Hospital/Hasbro Children's Hospital.

DETAILED DESCRIPTION:
The clinical course of sickle cell disease (SCD) is very variable. Some patients experience vaso-occlusive disease infrequently, but other patients develop the complication recurrently. The reason for the difference remains unclear. Although erythrocyte sickling occurs due to factors such as dehydration, infections, extreme of temperatures, acidosis, and hypoxia, neutrophil adhesion and activation are crucial in eliciting the vaso-occlusive crisis in patients with SCD. Activated neutrophils upregulate the expression of various cellular adhesion molecules that increase their "stickiness" in vivo. A murine model of SCD demonstrated the importance of the intestinal microbiome in influencing the kinetics of ageing neutrophils. Depletion of the microbiota with prolonged courses of broad-spectrum systemic antibiotics resulted in a reduction of the number of these neutrophils and protection against LPS-induced fatal vaso-occlusive crisis in these mice.

Intestinal barrier is a functional barrier that separates the gut lumen from the inner host. It consists of mechanical elements (mucus, epithelial layer), humoral elements (defensins, IgA), immunologic elements (lymphocytes, innate immune cells), muscular and neurological element. Although the normal intestinal microbiota is the main source of endogenous pathogens, it also contributes to the functional integrity of the intestinal barrier through its interaction with the other components of the barrier. Failure of any of these components will result in a breakdown of the protective intestinal barrier with the consequence of recurrent intestinal-derived bacteremia/septicemia. A breakdown of the normal microbiome has been implicated in the development of various pathologic states, including Clostridium difficile infection, inflammatory bowel disease, intestinal graft-versus-host disease following allogeneic hematopoietic progenitor cell transplant, colon cancer, and metabolic disorders such as obesity and non-alcoholic steatohepatitis.

To explain the reason for the development of frequent vaso-occlusive crisis in some patients with SCD, the investigators' stepwise hypothesis is that, due to the sickling process and the consequent development of intestinal ischemia, patients with SCD, especially those with frequent vaso-occlusive crisis, are more likely to have altered microbiota than healthy individuals. If the normal microbiota is altered, the intestinal barrier will be compromised, rendering the patients more susceptible to recurrent bacteremia of intestinal origin. Since most SCD patients with vaso-occlusive crisis present without any obvious infections, it is likely that the compromised intestinal barrier facilitates an inoculum of bacteremia not high enough to cause overt infections but sufficient to activate neutrophils and elicit vaso-occlusive crisis. The first step towards testing this overall hypothesis is to test the sub-hypothesis that altered intestinal microbiomes correlate with increased number of activated neutrophils and frequent vaso-occlusive crisis in patients with SCD.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female will be accrued to the study, without any pre-specified sex ratio.
2. Subject must have either HbSS or HbS/beta thal.
3. Subject is >8 years of age; if subject is <18 years, parental consent is needed.
4. Understands the process of and is willing to provide a written consent.

Exclusion Criteria:

1. Is taking immunosuppressive agents, including corticosteroids with prednisone at a dose of > 30 mg/day or other forms of corticosteroid at the equivalent dose.
2. Has taken systemic antimicrobials (except prophylactic Penicillin) in the preceding two weeks.
3. Has had a vaso-occlusive crisis in the preceding two weeks.
4. Has a history of colon cancer or an inflammatory bowel disease.
5. Has a history of clostridium difficile infection in the preceding eight weeks.
6. History of psychiatric disorder which in the investigators opinion may compromise compliance with the protocol or which does not allow for appropriate informed consent.
7. Pregnant or lactating females.
8. Patients who are court-mandated to reside at a treatment facility (e.g., drug or psychiatric treatment) or prison.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with SCD attending the hematology clinic at Rhode Island Hospital will be invited to participate in this study. A total of 50 eligible patients will be accrued to the study. Participation in the study is voluntary and the subject will not receive any compensation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Fecal microbiome | 1 year

IPD SHARING:
Plan to Share IPD: No